CLINICAL TRIAL: NCT06073210
Title: Mental Practice and Therapeutic Exercise in Young Nulliparous Women: A Randomized Controlled Trial
Brief Title: Mental Practice and Therapeutic Exercise in Young Nulliparous Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Ferran Cuenca, PhD, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UV0001
Record Dates: First submitted 2023-10-03; First posted 2023-10-10 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Therapeutic Exercise; Motor Imagery; Action Observation
MeSH Terms: interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Therapeutic exercise plus motor imagery (Experimental): This group will perform a therapeutic exercise programme (aerobic and strength training) to which motor imagery training will be added.
  Interventions: Behavioral: Motor Imagery plus therapeutic exercise
- Therapeutic exercise plus action observation (Experimental): This group will perform a therapeutic exercise programme (aerobic and strength training) to which action observation training will be added.
  Interventions: Behavioral: Action observation plus therapeutic exercise
- Therapeutic exercise (Active Comparator): This group will perform a therapeutic exercise programme (aerobic and strength training) to which sham action observation training will be added.
  Interventions: Behavioral: Sham action observation plus therapeutic exercise

INTERVENTIONS:
Behavioral: Motor Imagery plus therapeutic exercise — Aerobic exercise (20 minutes) and strengthening exercise (15 minutes) to which will be added a motor imagery intervention (imagining movements without actually doing them).
  Arms: Therapeutic exercise plus motor imagery
Behavioral: Action observation plus therapeutic exercise — Aerobic exercise (20 minutes) and strengthening exercise (15 minutes) to which will be added a action observation intervention (observing movements without actually doing them).
  Arms: Therapeutic exercise plus action observation
Behavioral: Sham action observation plus therapeutic exercise — Aerobic exercise (20 minutes) and strengthening exercise (15 minutes) to which will be added a sham action observation intervention (observing space planets).
  Arms: Therapeutic exercise

SUMMARY:
Mental practice (both in isolation and also in combination with real practice) has been shown to improve somatosensory and motor variables but so far no study has taken it into the study of women's health. Through this study we want to offer some interesting data regarding the effectiveness of mental practice combined with physical practice.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years of age and asymptomatic women.

Exclusion Criteria:

* This study will exclude those who presented a respiratory pathology, cardiac, systematic, or metabolic disease, history of recent surgery, vertebral fracture, or osteoarticular disorders of the spine area.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-09-30 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Pelvic Floor Muscle Strength | pre-intervention (T0), and inmmediate post-intervention (T1) (between the first and the second measurement, about 60 minutes have elapsed because it is done on the same day).
  maximum pelvic floor strength
Pain Pressure Threshold | pre-intervention (T0), and inmmediate post-intervention (T1) (between the first and the second measurement, about 60 minutes have elapsed because it is done on the same day).
  Pain sensitivity
Lumbopelvic Motor Control | pre-intervention (T0), and inmmediate post-intervention (T1) (between the first and the second measurement, about 60 minutes have elapsed because it is done on the same day).
  Sensorimotor control of lower limbs

CONTACTS AND LOCATIONS:
Locations (1):
- Ferran Cuenca Martínez, Valencia, Spain